CLINICAL TRIAL: NCT06939621
Title: Trajectories for Active and Healthy Aging (Behavioural and Psychological Determinants)
Brief Title: Trajectories for Active and Healthy Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Andrea Chirico, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CERT_1908372DCC2
Record Dates: First submitted 2025-03-18; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Older Adults (65 Years and Older); Virtual Reality; Physical Activity
Keywords: Older adult; Virtual Reality; Physical Activity; Self-Determination Theory; Motivation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial, including 60 older adults, were divided into four groups each involved in a 4 week intervention under 4 different conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental Group 1: VR-based intervention with motivational messages (Active Comparator): Participants will receive a VR-based physical exercise intervention featuring a virtual coach (an older adult peer) who provides both instructions and motivational messages based on Self-Determination Theory (SDT) during the session.
  Interventions: Behavioral: VR-based physical activity with motivational stimuli
- Experimental Group 2: VR-based intervention without motivational messages (Active Comparator): Participants will receive a VR-based physical exercise intervention featuring a virtual coach (an older adult peer) who provides both instructions and informative messages during the session.
  Interventions: Behavioral: VR-based physical activity without motivational stimuli
- Control Group 1: standard physical activity intervention with motivational messages (Active Comparator): Participants will take part in a standard physical activity intervention led by a real coach who provides both instructions and motivational messages based on SDT.
  Interventions: Behavioral: Standard Physical Activity with motivational stimuli
- Control Group 2: standard physical activity intervention without motivational messages (Active Comparator): Participants will take part in a standard physical activity intervention led by a real coach who provides both instructions and informative messages.
  Interventions: Behavioral: Standard Physical Activity without motivational stimuli

INTERVENTIONS:
Behavioral: VR-based physical activity with motivational stimuli — Participants will undergo four weekly supervised VR-based training sessions, each lasting approximately 35 minutes, over four weeks. Each session includes:
  1. VR Warm-Up: Activities adapted from NVIDIA VR Fun House on SteamVR, involving repetitive movements through mini-games like throwing objects, archery, and sword handling.
  2. Aerobic and Balance Exercises: Walking in place within a virtual natural environment, incorporating stretching steps and one-leg balance tasks.
  3. Lower-Body Training: VR-based exercises such as Balloon Game for hip flexibility (popping balloons with foot movements), Cave Game for squatting motions, and sit-to-stand activities.
  4. Upper-Body Training: VR exercises involving racket-based ball hitting and reaching activities at varied distances.
  Participants received motivational messages from a virtual coach designed to enhance the three psychological needs outlined in Self-Determination Theory: competence, autonomy, and relatedness.
  Arms: Experimental Group 1: VR-based intervention with motivational messages
Behavioral: VR-based physical activity without motivational stimuli — Participants will undergo four weekly supervised VR-based training sessions, each lasting approximately 35 minutes, over four weeks. Each session includes:
  1. VR Warm-Up: Activities adapted from NVIDIA VR Fun House on SteamVR, involving repetitive movements through mini-games like throwing objects, archery, and sword handling.
  2. Aerobic and Balance Exercises: Walking in place within a virtual natural environment, incorporating stretching steps and one-leg balance tasks.
  3. Lower-Body Training: VR-based exercises such as Balloon Game for hip flexibility (popping balloons with foot movements), Cave Game for squatting motions, and sit-to-stand activities.
  4. Upper-Body Training: VR exercises involving racket-based ball hitting and reaching activities at varied distances.
  In this condition, instead of motivational stimuli, participants received neutral information regarding the activity (e.g., "This exercise is good for your legs ").
  Arms: Experimental Group 2: VR-based intervention without motivational messages
Behavioral: Standard Physical Activity with motivational stimuli — Participants will engage in four individual training sessions, supervised by a trainer, scheduled once per week for a total duration of four weeks. Each session will last approximately 35 minutes and include: 5 minutes of warm-up and stretching, 10 minutes of aerobic and balance exercises (walking in place, heel raises, knee lifts, leg curls), 10 minutes of lower-body exercises (squats), and 10 minutes of upper-body exercises (shoulder abduction 180°, shoulder flexion 180°, shoulder external rotation 90°, bending 35°, trunk extensions 80°).
  Participants received motivational messages from a real coach designed to enhance the three psychological needs outlined in Self-Determination Theory: competence, autonomy, and relatedness.
  Arms: Control Group 1: standard physical activity intervention with motivational messages
Behavioral: Standard Physical Activity without motivational stimuli — Participants will engage in four individual training sessions, supervised by a trainer, scheduled once per week for a total duration of four weeks. Each session will last approximately 35 minutes and include: 5 minutes of warm-up and stretching, 10 minutes of aerobic and balance exercises (walking in place, heel raises, knee lifts, leg curls), 10 minutes of lower-body exercises (squats), and 10 minutes of upper-body exercises (shoulder abduction 180°, shoulder flexion 180°, shoulder external rotation 90°, bending 35°, trunk extensions 80°). In this condition, instead of motivational stimuli, participants received neutral information regarding the activity (e.g., "This exercise is good for your legs ").
  Arms: Control Group 2: standard physical activity intervention without motivational messages

SUMMARY:
The objective of the present study is to identify which psychological and motivational factors can help foster Virtual Reality (VR)-based interventions. Specifically, the main question is:

- Does the combination of VR-based interventions and motivational messages grounded in Self-Determination Theory (SDT) impact older adults' motivation for physical activity and their physiological indicators related to exercise? Older adults will participate to a 4 week intervention where they have ti engage in a physical activity program under different conditions: with and without VR, with and with out motivational messages.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years old
* to be fluent in Italian
* to have an informant familiar with their daily functioning
* needed to be available for the full duration of the study
* to be free from a history of severe psychiatric disorders (e.g., schizophrenia, bipolar disorder), nervous system infections or disorders (e.g., epilepsy, brain tumor, large-vessel stroke, major head trauma), or current metabolic or systemic conditions (e.g., B12 deficiency, renal failure, cancer)

Exclusion Criteria:

* severe sensory or motor impairments that would hinder task performance (e.g., blindness, total hearing loss, severe upper extremity deformities or paralysis)
* susceptibility to motion sickness (as confirmed by the Motion Sickness Susceptibility Questionnaire)
* intellectual disability (as assessed by the MMSE).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Physical activity | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  The Godin-Shephard Leisure-Time Physical Activity Questionnaire. The GSLTPAQ comprises three items, each representing a different intensity of exercise: strenuous (e.g., running), moderate (e.g., fast walking), and mild (e.g., yoga). Participants report the number of times per week they engage in 20 minutes of strenuous, moderate, and mild exercise during their free time. To calculate the Leisure Score Index (LSI), the weekly duration of each activity type is multiplied by its respective Metabolic Equivalent Task (MET) value: 3 for mild, 5 for moderate, and 9 for strenuous. Larger values indicate higher levels of engagement in physical activity.
Basic Psychological Needs | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  The Psychological Need Satisfaction in Exercise Scale (PNSE) was used to assess SDT basic psychological needs. The PNSE consists of 18 items, rated on a 6-point Likert scale (from 1 ="false" to 6 = "true"). Larger values indicate higher satisfaction of basic psychological needs.
Motivation for physical activity | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  The Behavioural Regulations in Exercise Questionnaire (BREQ-3) was use to assess motivation for physical activity as poised by the Self-Determination Theory. It consists of 18 items rated on a five-point Likert scale, ranging from 0 ("not true for me") to 4 ("very true for me").
General Physical Health | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  Physical health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better physical health.
General Mental Health | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  Mental health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better mental health.
Physiological measures of Physical Activity: Hearth rate variability | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  Hearth rate variability was measure through the smartwatch EMPATICA EmbracePlus.
Physiological measures of Physical Activity: galvanic conductance | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  Galvanic conductance was measure through the smartwatch EMPATICA EmbracePlus.
Physical activity | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  The Godin-Shephard Leisure-Time Physical Activity Questionnaire. The GSLTPAQ comprises three items, each representing a different intensity of exercise: strenuous (e.g., running), moderate (e.g., fast walking), and mild (e.g., yoga). Participants report the number of times per week they engage in 20 minutes of strenuous, moderate, and mild exercise during their free time. To calculate the Leisure Score Index (LSI), the weekly duration of each activity type is multiplied by its respective Metabolic Equivalent Task (MET) value: 3 for mild, 5 for moderate, and 9 for strenuous. Larger values indicate higher levels of engagement in physical activity.
Basic Psychological Needs | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  The Psychological Need Satisfaction in Exercise Scale (PNSE) was used to assess SDT basic psychological needs. The PNSE consists of 18 items, rated on a 6-point Likert scale (from 1 ="false" to 6 = "true"). Larger values indicate higher satisfaction of basic psychological needs.
Motivation for physical activity | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  The Behavioural Regulations in Exercise Questionnaire (BREQ-3) was use to assess motivation for physical activity as poised by the Self-Determination Theory. It consists of 18 items rated on a five-point Likert scale, ranging from 0 ("not true for me") to 4 ("very true for me").
General Physical Health | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  Physical health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better physical health.
General Mental Health | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  Mental health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better mental health.
Physiological measures of Physical Activity: hearth rate variability | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  Hearth rate variability was measure through the smartwatch EMPATICA EmbracePlus.
Physiological measures of Physical Activity: galvanic conductance | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  Galvanic conductance was measure through the smartwatch EMPATICA EmbracePlus.
Physical activity | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  The Godin-Shephard Leisure-Time Physical Activity Questionnaire. The GSLTPAQ comprises three items, each representing a different intensity of exercise: strenuous (e.g., running), moderate (e.g., fast walking), and mild (e.g., yoga). Participants report the number of times per week they engage in 20 minutes of strenuous, moderate, and mild exercise during their free time. To calculate the Leisure Score Index (LSI), the weekly duration of each activity type is multiplied by its respective Metabolic Equivalent Task (MET) value: 3 for mild, 5 for moderate, and 9 for strenuous. Larger values indicate higher levels of engagement in physical activity.
Basic Psychological Needs | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  The Psychological Need Satisfaction in Exercise Scale (PNSE) was used to assess SDT basic psychological needs. The PNSE consists of 18 items, rated on a 6-point Likert scale (from 1 ="false" to 6 = "true"). Larger values indicate higher satisfaction of basic psychological needs.
Motivation for physical activity | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  The Behavioural Regulations in Exercise Questionnaire (BREQ-3) was use to assess motivation for physical activity as poised by the Self-Determination Theory. It consists of 18 items rated on a five-point Likert scale, ranging from 0 ("not true for me") to 4 ("very true for me").
General Physical Health | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  Physical health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better physical health.
General Mental Health | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  Mental health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better mental health.
Physiological measures of Physical Activity: hearth rate variability | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  Hearth rate variability was measure through the smartwatch EMPATICA EmbracePlus.
Physiological measures of Physical Activity: galvanic conductance | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  Galvanic conductance was measure through the smartwatch EMPATICA EmbracePlus.
Physical activity | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  The Godin-Shephard Leisure-Time Physical Activity Questionnaire. The GSLTPAQ comprises three items, each representing a different intensity of exercise: strenuous (e.g., running), moderate (e.g., fast walking), and mild (e.g., yoga). Participants report the number of times per week they engage in 20 minutes of strenuous, moderate, and mild exercise during their free time. To calculate the Leisure Score Index (LSI), the weekly duration of each activity type is multiplied by its respective Metabolic Equivalent Task (MET) value: 3 for mild, 5 for moderate, and 9 for strenuous. Larger values indicate higher levels of engagement in physical activity.
Basic Psychological Needs | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  The Psychological Need Satisfaction in Exercise Scale (PNSE) was used to assess SDT basic psychological needs. The PNSE consists of 18 items, rated on a 6-point Likert scale (from 1 ="false" to 6 = "true"). Larger values indicate higher satisfaction of basic psychological needs.
Motivation for physical activity | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  The Behavioural Regulations in Exercise Questionnaire (BREQ-3) was use to assess motivation for physical activity as poised by the Self-Determination Theory. It consists of 18 items rated on a five-point Likert scale, ranging from 0 ("not true for me") to 4 ("very true for me").
General Physical Health | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  Physical health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better physical health.
General Mental Health | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  Mental health was assessed using the 12-Item Short Form Survey (SF-12), which comprises 12 items. Raw scores are transformed into T-scores, with higher scores indicating better mental health.
Physiological measures of Physical Activity: galvanic conductance | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  Galvanic conductance was measure through the smartwatch EMPATICA EmbracePlus.
Physiological measures of Physical Activity: hearth rate variability | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  Hearth rate variability was measure through the smartwatch EMPATICA EmbracePlus.

SECONDARY OUTCOMES:
Well-being | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  The Subjective Vitality/Depletion Scale was use to assess well-being. This self-report questionnaire is composed of six items rated on a 7-point Likert scale (from 1 = "Not at all true" to 7 = "Very true"). Higher scores are indicative of higher well-being.
Self-Efficacy for exercise | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  The Self-Efficacy for Exercise Scale (SEE) is a self-report questionnaire composed of nine items for the assessment of self-efficacy for exercise, specifically designed for older adults. Each item is rated on an 11-point scale (from 0 = "Not confident" to 10 = "Very confident"). Scores ranges from a minimum of 0 to a maximum of 90. Larger values reflects higher degree of confidence that an elder has in engaging in exercise in the presence of specific barriers.
Virtual reality experience: physical symptoms | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for physical symptoms range from 0 to 48. Higher scores indicate greater discomfort.
Virtual reality experience: eye-related symptoms | Week 1, day 1 (Exercise session 1). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for eye-related symptoms range from 0 to 40. Higher scores indicate greater discomfort.
Well-being | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  The Subjective Vitality/Depletion Scale was use to assess well-being. This self-report questionnaire is composed of six items rated on a 7-point Likert scale (from 1 = "Not at all true" to 7 = "Very true"). Higher scores are indicative of higher well-being.
Self-Efficacy for exercise | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  The Self-Efficacy for Exercise Scale (SEE) is a self-report questionnaire composed of nine items for the assessment of self-efficacy for exercise, specifically designed for older adults. Each item is rated on an 11-point scale (from 0 = "Not confident" to 10 = "Very confident"). Scores ranges from a minimum of 0 to a maximum of 90. Larger values reflects higher degree of confidence that an elder has in engaging in exercise in the presence of specific barriers.
Virtual reality experience: physical symptoms | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for physical symptoms range from 0 to 48. Higher scores indicate greater discomfort.
Virtual reality experience: eye-related symptoms | Week 2, day 2 (Exercise session 2). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for eye-related symptoms range from 0 to 40. Higher scores indicate greater discomfort.
Well-being | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  The Subjective Vitality/Depletion Scale was use to assess well-being. This self-report questionnaire is composed of six items rated on a 7-point Likert scale (from 1 = "Not at all true" to 7 = "Very true"). Higher scores are indicative of higher well-being.
Self-Efficacy for exercise | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  The Self-Efficacy for Exercise Scale (SEE) is a self-report questionnaire composed of nine items for the assessment of self-efficacy for exercise, specifically designed for older adults. Each item is rated on an 11-point scale (from 0 = "Not confident" to 10 = "Very confident"). Scores ranges from a minimum of 0 to a maximum of 90. Larger values reflects higher degree of confidence that an elder has in engaging in exercise in the presence of specific barriers.
Virtual reality experience: physical symptoms | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for physical symptoms range from 0 to 48. Higher scores indicate greater discomfort.
Virtual reality experience: eye-related symptoms | Week 3, day 3 (Exercise session 3). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for eye-related symptoms range from 0 to 40. Higher scores indicate greater discomfort.
Well-being | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  The Subjective Vitality/Depletion Scale was use to assess well-being. This self-report questionnaire is composed of six items rated on a 7-point Likert scale (from 1 = "Not at all true" to 7 = "Very true"). Higher scores are indicative of higher well-being.
Self-Efficacy for exercise | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  The Self-Efficacy for Exercise Scale (SEE) is a self-report questionnaire composed of nine items for the assessment of self-efficacy for exercise, specifically designed for older adults. Each item is rated on an 11-point scale (from 0 = "Not confident" to 10 = "Very confident"). Scores ranges from a minimum of 0 to a maximum of 90. Larger values reflects higher degree of confidence that an elder has in engaging in exercise in the presence of specific barriers.
Virtual reality experience: physical symptoms | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for physical symptoms range from 0 to 48. Higher scores indicate greater discomfort.
Virtual reality experience: eye-related symptoms | Week 4, day 4 (Exercise session 4). The measurement will take place after and before the exercise session.
  Virtual Reality Symptoms Questionnaire. This self-report questionnaire comprises 13 items divided into two dimensions: physical symptoms (8 items) and eye-related symptoms (5 items). Each item is rated on a 7-point Likert scale (ranging from 0 = "none" to 6 = "severe"). Scores for eye-related symptoms range from 0 to 40. Higher scores indicate greater discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Lucidi, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No